CLINICAL TRIAL: NCT03157271
Title: The Addition of Dry Needling in the Treatment of Patients With Patellofemoral Pain Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00081677
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-08

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFPS Treatment (No Intervention): This arm (group of patients) will receive typical/pragmatically designed treatment for patellofemoral pain syndrome.
- PFPS Plus Dry Needling Treatment (Experimental): This group will receive the same typical/pragmatically designed treatment for patellofemoral pain syndrome but with the addition of a dry needling intervention.
  Interventions: Other: Intramuscular Dry Needling

INTERVENTIONS:
Other: Intramuscular Dry Needling — Dry Needling is a procedure in which a solid filament needle is inserted into the skin and muscle directly at a myofascial trigger point. A myofascial trigger point consists of multiple contraction knots, which are related to the production and maintenance of the pain cycle and interfere with movement patterns.
  Other Names: Trigger Point Dry Needling
  Arms: PFPS Plus Dry Needling Treatment

SUMMARY:
Subjects between 14 and 40 years of age referred to physical therapy with a diagnosis of PFPS will be randomly assigned to one of two groups. The first group (PFPS) will be treated pragmatically. The second group (PFPS+DN) will receive the same pragmatic approach with the addition of dry needling intervention. The dry needling intervention will be delivered based on the treating physical therapist's examination of the patient's soft tissue mobility deficits, muscle activation deficits, or referred pain patterns.

DETAILED DESCRIPTION:
All interventions delivered to both study groups will be provided by licensed physical therapists at Duke Sports Medicine. The frequency of visits and duration of physical therapy care will be determined on an individual basis. Both groups will be expected to perform an individualized home exercise program to supplement formal therapy visits. The PFPS group will receive a pragmatic treatment approach reflective of currently accepted interventions. The clinician will have the ability to select appropriate interventions based on the presentation/need of each patient. These interventions may include: stretching (iliotibial band, hip flexor, lateral retinaculum); patellar taping; kinesiology taping; bracing; joint mobilization (patella, ankle, hip); orthotics/footwear recommendations; pain modalities such as Ice, electric stimulation, laser; soft tissue mobilization (manual or instrument assisted) for restricted tissues such as peri-patellar tissues, iliotibial band, tensor fasciae latae, hamstrings, calf, quadriceps, hip flexors, and gluteals. The PFPS+DN group will be treated in the same manner described above with the addition of the dry needling intervention. The dry needling intervention will be prescriptive in that each provider will assess patient for the presence of a trigger point that may be contributing either directly or indirectly to the patient's symptoms and perform the intervention per the following guidelines. First, the presence of a trigger point must be verified by locating a palpable taught band, a hypersensitive tender area, referred pain of the MTrP in response to compression, a Jump Sign - response from patient who winces, may cry out, or withdraw, or a local twitch response provoked by manually snapping the taut band. Second, a muscle may be selected for dry needling if that muscle is assumed to be contributing to tissue extensibility restriction, motor control dysfunction, or hyperactivity.

ELIGIBILITY:
Inclusion Criteria:

* Anterior or retro-patellar knee pain from at least two of the following: prolonged sitting, stair climbing, squatting, running, kneeling, and hopping/jumping.
* Insidious onset of symptoms unrelated to trauma
* Presence of pain on palpation of the patellar facets
* Pain on compression of the patella

Exclusion Criteria:

* Signs or symptoms of meniscal or other intra-articular pathologic condition.
* Self-reported other knee pathology such as cartilage injury or ligamentous tear.
* Known articular cartilage damage (from previously obtained imaging).
* Ligament laxity or tenderness.
* Patellar tendonitis, ITB syndrome, fracture,
* Tenderness over the patellar tendon, ITB, tibial tubercle, or pes anserinus tendons "if reproduced the pain"
* Patellar instability (positive apprehension sign and/or self-reported history of dislocations or subluxations.
* Concurrent Hip Pain
* Lumbar referred pain
* Osgood-Schlatters or Sinding-Larsen-Johanssen Syndromes
* Knee surgery within the past year
* Evidence of effusion

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in Lower Extremity Functional Scale | Baseline, 2 weeks, 1 month, at completion of treatment (average of 10 weeks), 3 months, 6 months
  20 Item Survey - Self report of difficulty with 20 lower extremity common tasks

SECONDARY OUTCOMES:
Change in Pain | Baseline, Days 1-15, 1 month, at completion of treatment (average of 10 weeks), 3 months, 6 months
  Subjective Report of Pain on a Scale from 0-10
Change in Global Function Rating | Baseline, Days 1-15, 1 month, at completion of treatment (average of 10 weeks), 3 months, 6 months
  Subjective Rating for Physical Function on a Scale from 0-100%
Change in Global Rating of Change | Baseline, Days 1-15, 1 month, at completion of treatment (average of 10 weeks), 3 months, 6 months
  Subjective Rating of Change since starting treatment scale of -7 (much worse) to +7 (much better)

IPD SHARING:
Plan to Share IPD: No